CLINICAL TRIAL: NCT00177086
Title: Alfuzosin Hydrochloride to Promote Passage of Distal Ureteral Calculi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Manoj, Monga, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0412M65851; L9839; 3579B
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Kidney Calculi; Ureteral Calculi; Colic
MeSH Terms: conditions — Kidney Calculi; Ureteral Calculi; Colic | interventions — alfuzosin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alfuzosin (Experimental)
  Interventions: Other: Alfuzosin Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Other: Alfuzosin Hydrochloride

INTERVENTIONS:
Other: Alfuzosin Hydrochloride — One tablet every day for 4 weeks
  Other Names: Sugar pill

SUMMARY:
This study will assess improvement in the percentage of spontaneous stone passage for distal ureteral calculi for alfuzosin compared to placebo, decrease of pain and narcotic/analgesic use associated with stone passage, decrease of the time to spontaneous stone passage, shift in the size distribution of stones passed towards larger sizes.

ELIGIBILITY:
Inclusion Criteria:

* Age =>18
* <8mm ureteral calculus below the pelvic brim identified by non-contrast CT scan and/or intravenous pyelogram

Exclusion Criteria:

* Subject with know hypersensitivity to Alfuzosin hydrochloride or any component of Alfuzosin hydrochloride tablets
* Pregnant/Nursing females
* Solitary kidney
* Renal insufficiency (Creatinine>1.8)
* Urinary infection (fever >101, positive urine culture, many bacteria on urinalysis)
* Moderate or severe hepatic insufficiency (Childs-Pugh categories B and C)
* Potent CYP3A4 inhibitors such as ketoconazole, itraconazole, and ritonavir, since Alfuzosin blood levels are increased
* Other alpha-blockers
* Phosphodiesterase type 5 inhibitors for erectile dysfunction
* Any subject for whom the principal investigator feels it would not be in his or her best interest to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Spontaneous stone passage for distal ureteral calculi | increased

SECONDARY OUTCOMES:
Decrease the pain and narcotic use associated with stone passage | decrease
Decrease the time to spontaneous passage | decrease
Shift the size distribution of stones passed towards larger sizes

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Monga, MD, Principal Investigator — University of Minnesota and VAMC Minneapolis
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States